CLINICAL TRIAL: NCT04682067
Title: Incentives to Promote Smoking Cessation for Individuals With Diabetes
Brief Title: Diabetes Smoking Cessation Incentives Study
Acronym: CRUK2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11582
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Smoking Cessation; Diabetes Type 2
Keywords: financial incentives; contingency management
MeSH Terms: conditions — Smoking Cessation; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency Management (Experimental): Participants in the contingency management (CM) treatment arm will receive the usual care (UC) treatment program offered at the Tobacco Treatment Research Program (TTRP) and will be eligible to earn gift cards at each weekly visit on their quit date up until four weeks post-quit for proof of abstinence. They will earn $20 in gift cards for quitting on the specified quit day (i.e., one week after the orientation visit), and this amount will increase by $5 with each successive weekly abstinent visit (i.e., up to $40 in gift cards at 4 weeks post-quit; up to $150 total).
  Interventions: Behavioral: Contingency Management; Behavioral: Usual Care smoking cessation
- Usual Care (Placebo Comparator): Participants in the usual care (UC) group will receive the standard smoking cessation treatment offered at the Health Promotion Research Center's Tobacco Treatment Research Program (TTRP) at the University of Oklahoma. This includes at least 4 treatment sessions of counseling and the opportunity to use nicotine replacement therapy or medications.
  Interventions: Behavioral: Usual Care smoking cessation

INTERVENTIONS:
Behavioral: Contingency Management — Escalating financial incentives contingent upon biochemical evidence of abstinence
  Arms: Contingency Management
Behavioral: Usual Care smoking cessation — Usual care smoking cessation support

SUMMARY:
The purpose of this study is to evaluate the feasibility of contingency management on improving smoking cessation among individuals with type 2 diabetes.

DETAILED DESCRIPTION:
Type 2 diabetes (T2DM) and cigarette smoking are major causes of morbidity and mortality in US, and research indicates there is a complex relationship between these two risk factors. Smoking cessation is recommended as a standard treatment of diabetes by the American Diabetes Association; however, patients with T2DM and their providers are often inundated with other challenging lifestyle changes and disease management. Due to the complex relationship between diabetes and smoking and the large number of competing lifestyle changes recommended at diagnosis, smokers with T2DM may benefit from a contingency management (CM) program that incentivizes cessation. Providing patients tangible rewards to reinforce positive behaviors such as smoking abstinence has been proven effective in substance abuse programs, smoking cessation among pregnant women unwilling or unable to quit, and other population subgroups. In this CRUK2 study the investigators aim to test and further explore the potential effectiveness of financial incentives contingent upon proof of quitting smoking. The investigators will gather diabetes-related contextual factors associated with participation in the program and smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* earn a score > 4 on REALM indicating > 6th grade English literacy level
* willing to quit smoking 7 days from their first visit
* have an expired CO level >8 ppm suggestive of current smoking at baseline
* currently smoking > 5 cigarettes per day
* willing and able to attend 6 study visits

Exclusion Criteria:

* unable to demonstrate use of or unwilling to use the remote CO monitor and phone app

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study has no inclusion/exclusion criteria based on gender
Enrollment: 29 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Number of participants completing 6 study visits | 5 weeks
  Feasibility outcome: completion of 6 study visits
Number of participants with >80% completion of daily ecological momentary assessments (EMA) completed | 4 weeks
  Feasibility outcome: completion of EMA portion of study

SECONDARY OUTCOMES:
Number of participants with biochemically verified abstinence at 4 weeks post quit | 5 weeks
  Carbon Monoxide (CO) ≤ 6 ppm on exit date; self-reported 7-day point prevalence abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Martinez, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Oklahoma Tobacco Research Center, Oklahoma City, Oklahoma, United States